CLINICAL TRIAL: NCT05360914
Title: Improving and Evaluation of a New Cross-sectoral Hospital at Home Model for Elderly Acute Ill Patients
Brief Title: Hospital at Home for Elderly Acute Ill Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Defactum, Central Denmark Region (Other Government)
Collaborators: Interdisciplinary Centre for Organizational Architecture (ICOA), Aarhus University, Denmark (Unknown); Research Center for Emergency Medicine, Aarhus University, Denmark (Unknown); Viborg Regional Hospital (Other)
Responsible Party: Principal Investigator, Camilla Palmhøj Nielsen, Research director, Defactum, Central Denmark Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Hospital at Home
Record Dates: First submitted 2022-04-21; First posted 2022-05-04 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cystitis; Erysipelas; Pneumonia
MeSH Terms: conditions — Cystitis; Erysipelas; Pneumonia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital at Home (HaH) treatment (Experimental): The patients in this arm will receive the intervention.
  Interventions: Other: Hospital at Home (HaH) treatment
- Standard hospital admission (Active Comparator): The patients in this arm are the control group and will receive the standard hospital treatment.
  Interventions: Other: Standard hospital admission

INTERVENTIONS:
Other: Hospital at Home (HaH) treatment — The intervention is a new pathway of providing acut treatment for elderly acute ill patients in their own home. If the patient is randomized to the intervention group, the municipalities acute teams start the treatment. The acute team can take venous blood tests, ECG and bladder scan at home. The acute team handles the treatment at home and follows the patient closely. During the treatment course, the acute team and the ED specialist discuss the treatment process either over the phone or virtually on an iPad, where the patient is also involved. If the specialist would like to see the patient for assessment or send the patient for an X-ray, the specialist informs the acute team that the patient must go to a short check-up in the ED. Here, the specialist examines the patient himself and assesses whether the patient can continue to be treated at home, or whether the patient must be admitted to the hospital due to deterioration of the condition.
  Arms: Hospital at Home (HaH) treatment
Other: Standard hospital admission — The active comparator is the standard hospital admission for elderly acute ill patients.
  Arms: Standard hospital admission

SUMMARY:
Many elderly patients with uncomplicated treatment courses are admitted unnecessarily, which is a burden for the patient and society. Studies show that Hospital at Home (HaH) treatment is an alternative to hospitalization. The patient's risk of delirium, infection and loss of function is reduced when the patient avoids the hospital stay. HaH treatment is expected to be more cost-effective, improve patients' functional abilities and patients' satisfaction.

Three municipalities, general practitioners, pre-hospital service and an emergency department (ED) in Central Denmark Region have organized the first HaH treatment model across disciplines and sectors. Specialists in the ED and the municipal acute teams provide HaH treatment for elderly acute ill patients. However, the model has not yet been evaluated.

The aim of this study is to optimize the HaH treatment model for elderly acute ill patients. The objective is to increase patient satisfaction and optimize the use of resources in healthcare by avoiding unnecessary hospitalizations that impair and prolong treatment.

This study is an open label randomized controlled trial (RCT) with a 1:2 allocation ratio of acute hospital admission versus HaH. During a pilot period, we tested and adapted the patient pathway of HaH to the practical reality, before we start the randomization for the RCT study. We will investigate the clinical effects and health economic consequences of HaH treatment compared with standard hospital treatment.

DETAILED DESCRIPTION:
Background

The Danish population that is above 65 years of age is expected to increase from 16% today to 25% in 2042. This will result in a larger demand for health care services, which is a task that the Danish hospital sector cannot perform alone. Emergency hospital admissions are not the best solution for treatment of all patients. For elderly, frail citizens an emergency admission is a big change in the daily life and often means a great risk of infection and delirium and loss of functional ability which takes a long time to regain.

The group of elderly medical patients is a broad group that demand a coherent and cross-sectoral treatment. This patient group is often only hospitalized for a short period. The hospitalization of these patients with rather uncomplicated treatment could possibly have been prevented if the collaboration between hospital, general practitioners (GPs), pre-hospital service and municipalities had been improved further.

These complex challenges underscore the need to explore innovative solutions. An alternative model of care that internationally has been identified as a possible solution is the Hospital at Home (HaH) treatment model. This model offers active treatment of a condition that otherwise would have demanded emergency admission and can be performed over a shorter period of time in patients' own home. Studies have shown that it is better for elderly patients to be treated in-home, and that patients that are treated in own home are more satisfied with their continuity of care. Many of these services are adjusted for elderly patients, but the services can be organized in different ways, focusing on different categories of patients.

During the last four years, GPs, an emergency department (ED), pre-hospital service, three municipalities, as well as researchers have organized the first HaH treatment model for elderly acute ill patients in a Danish context, but it has not yet been implemented or evaluated. The aim of this study is to optimize the HaH treatment model for elderly acute ill patients. The objective is to increase patient satisfaction and optimize the use of resources in healthcare by avoiding unnecessary hospitalizations that impair and prolong treatment. We will investigate the clinical effects and health economic consequences of HaH treatment compared with standard hospital treatment using an open labelled RCT design.

Study design and setting

This study was approved by the Ethical Committee, Central Denmark Region (no. 1-10-72-67-20). To qualify the patient pathway and to ensure the generalizability, we will conduct an open labelled RCT with two arms in collaboration between GPs, three municipalities (Viborg, Skive and Silkeborg), pre-hospital service, ED at the Regional Hospital, Viborg in the period between June 1, 2022, and August 31, 2024. A steering group and a task force have been established, in which all organizational units that form part of the research project are represented and actively participating. Researchers affiliated DEFACTUM, Aarhus University, and Research Center for Emergency Medicine support the cross-sectoral collaboration. The study was designed in accordance with the SPIRIT 2013 statement (Standard Protocol Items: Recommendations for Interventional Trials).

Participants

Patients with an acute medical condition will be invited to participate in the study. Other inclusion criteria are:

* The patient should be aged 65 and over
* Diagnosed with a stable acute medical conditions e.g. cystitis, erysipelas, pneumonia
* The patient should be living in their own home or a nursing home before entering the study
* The patient should be residing in one of the three municipalities (Viborg, Skive and Silkeborg)
* The patient must have been seen by the GP in the case of disease in question
* The patient should speak and understand Danish.
* The patient should give informed consent to participate in the study.

Exclusion criteria are:

* The patient is unable to give written consent
* The capacity of the municipal acute team care was fully utilised.

Randomization

Patients will be identified by their GP or the referring physician (on-call or ambulance doctor). Then the GP or the referring physician (on-call or ambulance doctor) and an ED physician will jointly through a conference call evaluate whether the patient can be included in the study. The conference call is a medical assessment of the patient to ensure that patient has the criteria for the inclusion in the study.

The participating patients are randomized using REDCap to the intervention group or control group, which ensures random distribution of patients in the ratio 1: 2, so that the two groups of patients are comparable. The randomisation process will be performed by the hospital visitation at ED. The investigators, patients, GPs, pre-hospital service and the ED can not influence to which group the patients will be allocated to. The ED, GP, pre-hospital service, investigators and patients will not be masked to the allocation.

All patients included will receive an information booklet and get oral information about the research project. At the first visit of the acute team, the patient gets an information booklet and is informed orally about the project. Then, informed consent is obtained to get relevant information from electronic patient journal.

Intervention

If the patient is randomized to the intervention group, the municipalities acute teams start the treatment. The acute team can take venous blood tests, ECG and bladder scan at home. The acute team, which is available around the clock, handles the treatment at home and follows the patient closely. During the treatment course, the acute team and the ED specialist discuss the treatment process either over the phone or virtually on an iPad, where the patient is also involved. If the specialist would like to see the patient for assessment or send the patient for an X-ray, the specialist informs the acute team that the patient must go to a short check-up in the ED. Here, the specialist examines the patient himself and assesses whether the patient can continue to be treated at home, or whether the patient must be admitted to the hospital due to deterioration of the condition. The ED specialist is responsible for discharging the patient. If the patient is randomized to the control group, the patient will receive the standard hospital treatment.

Power calculations

An outcome in the project is the proportion of 30-days of acute hospitalization, which is an outcome that can support a power calculation for the project. Levine et al. shows that the proportion of 30-days acute hospitalization for patients who have been treated in their own home is 0.07, while for patients in the hospital it is 0.13. In order for us to show a difference in the proportion of acute readmissions with a significance level of 5% and 80% power and a ratio of 1: 2, there must be 283 patients in the control group and 566 patients in the intervention group. A total of 849 patients living in Viborg, Skive and Silkeborg Municipalities will be included in the study.

Data and statistical analysis

Data will be partly obtained from the Danish National Registries. Furthermore, data on resource use in HaH group, EuroQoL-5 Dimensions (EQ-5D) and the functional test Timed up and Go (TUG) will be be entered into dedicated databases and stored in accordance with the Danish Data Protection Agency requirements.

Statistical analyses will be based on 'intention to treat' principles and will be performed using STATA 16. Descriptive statistics will be conducted to describe baseline variables. Logistic regression will be used to analyse the binary outcomes and the continuous outcomes will be analysed using linear regression. The results will be reported in accordance with CONSORT 2010 statement.

ELIGIBILITY:
Inclusion Criteria:

* The patient should be aged 65 and over
* Diagnosed with a stable acute medical conditions e.g. cystitis, erysipelas, pneumonia
* The patient should be living in their own home or a nursing home before entering the study
* The patient should be residing in one of the three municipalities (Viborg, Skive and Silkeborg)
* The patient must have been seen by the GP or the pre-hospital service in the case of disease in question
* The patient should speak and understand Danish.
* The patient should give informed consent to participate in the study.

Exclusion Criteria:

* The patient is unable to give written consent
* The capacity of the municipal acut team care was fully utilised.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 849 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Rate of 30-days re-admission | 30 days period after discharge
  Rate of 30-days re-admission after discharge
Health Related Quality of Life | From inclusion to 3 months follow-up
  Estimating quality of life by using EuroQoL-5 Dimensions. We will use EuroQoL-5 Dimensions to measure Health Related Quality of Life. The five dimensions include mobility, self-care, usual activity, pain/discomfort and anexiety/depression.This tool will provide us with health states (11111 being the best health state and 55555 the worse health state). We will use the Danish weight to give weights to different health states obtained from EuroQoL-5 Dimensions.

SECONDARY OUTCOMES:
Functional mobility test | From inclusion to 3 months follow-up
  Estimating basic functional mobility by using Timed Up and Go (TUG)
Mortality rate | From inclusion to 3 months follow-up
  Estimating mortality rate for the study population using the National Registries
Number of contacts to primary and secondary health care system | From inclusion to 3 months follow-up
  The Danish National Registries will be used to estimate number of contacts to the primary and secondary healthcare for both control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Palmhøj Nielsen, Ph.D, Principal Investigator — Defactum, Central Denmark Region
Locations (3):
- Denmark (3):
  - Silkeborg municipality, Silkeborg
  - Skive municipality, Skive
  - Viborg municipality, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Creditor MC. Hazards of hospitalization of the elderly. Ann Intern Med. 1993 Feb 1;118(3):219-23. doi: 10.7326/0003-4819-118-3-199302010-00011. PMID 8417639
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Greenough WB 3rd, Guido S, Steinwachs D. Comparison of functional outcomes associated with hospital at home care and traditional acute hospital care. J Am Geriatr Soc. 2009 Feb;57(2):273-8. doi: 10.1111/j.1532-5415.2008.02103.x. Epub 2008 Dec 11. PMID 19170781
- [Background] Isaia G, Astengo MA, Tibaldi V, Zanocchi M, Bardelli B, Obialero R, Tizzani A, Bo M, Moiraghi C, Molaschi M, Ricauda NA. Delirium in elderly home-treated patients: a prospective study with 6-month follow-up. Age (Dordr). 2009 Jun;31(2):109-17. doi: 10.1007/s11357-009-9086-3. Epub 2009 Jan 30. PMID 19507055
- [Background] Wilson A, Wynn A, Parker H. Patient and carer satisfaction with 'hospital at home': quantitative and qualitative results from a randomised controlled trial. Br J Gen Pract. 2002 Jan;52(474):9-13. PMID 11791829
- [Background] Aimonino Ricauda N, Tibaldi V, Leff B, Scarafiotti C, Marinello R, Zanocchi M, Molaschi M. Substitutive "hospital at home" versus inpatient care for elderly patients with exacerbations of chronic obstructive pulmonary disease: a prospective randomized, controlled trial. J Am Geriatr Soc. 2008 Mar;56(3):493-500. doi: 10.1111/j.1532-5415.2007.01562.x. Epub 2008 Jan 4. PMID 18179503
- [Background] Shepperd S, Iliffe S. Hospital at home versus in-patient hospital care. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD000356. doi: 10.1002/14651858.CD000356.pub2. PMID 16034853
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Levine DM, Ouchi K, Blanchfield B, Saenz A, Burke K, Paz M, Diamond K, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: A Randomized Controlled Trial. Ann Intern Med. 2020 Jan 21;172(2):77-85. doi: 10.7326/M19-0600. Epub 2019 Dec 17. PMID 31842232
- [Background] Shepperd S, Doll H, Angus RM, Clarke MJ, Iliffe S, Kalra L, Ricauda NA, Wilson AD. Admission avoidance hospital at home. Cochrane Database Syst Rev. 2008 Oct 8;(4):CD007491. doi: 10.1002/14651858.CD007491. PMID 18843751
- [Derived] Thomsen AML, Tayyari N, Duvald I, Kirkegaard H, Obel B, Nielsen CP. Hospital at home for elderly acute patients: a study protocol for a randomised controlled trial. BMJ Open. 2024 May 2;14(5):e083372. doi: 10.1136/bmjopen-2023-083372. PMID 38697766
- See also: The Danish National program for elderly care — https://www.sst.dk/-/media/Udgivelser/2016/Styrket-indsats-for-den-aeldre-medicinske-patient.ashx?la=da&hash=8F69A91EB3B59BC7AF2ABA646A7089D99BCD660E
- See also: Effective municipality program with focus on prevention of admission and re-admission — https://sum.dk/Media/A/0/Effektiv-kommunal-forebyggelse.pdf